CLINICAL TRIAL: NCT02810210
Title: Études Observationnelles Des conséquences néonatales et pédiatriques de l'Infection à Virus Zika au Cours de la Grossesse Pendant l'épidémie Des départements français d'Amérique de l'année 2016
Brief Title: Zika Virus Infection's Neonatal and Pediatric Consequences in French Department of America
Acronym: ZIKA-DFA-BB
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-19
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Zika Virus Infection on Fetus and Child During the Pregnancy
Keywords: Zika; microcephaly; congenital abnormalities; new-born; infant
MeSH Terms: conditions — Zika Virus Infection; Microcephaly; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Monitoring of children born without congenital anomalies to mothers with biologically confirmed ZIKV's infection during the pregnancy
- Cohort 2: Monitoring of children born with congenital anomalies to mothers with biologically confirmed ZIKV's infection during the pregnancy
- Cohort 3: Monitoring of children born without congenital anomalies to mothers with no biologically confirmed ZIKV's infection during the pregnancy
  Interventions: Other: fundus examination; Other: Head ultrasound

INTERVENTIONS:
Other: fundus examination — In cohort 3, a fundus examination will be carried in addition to the current medical practice.
  This exam is part of current medical practice for other groups.
  Groups: Cohort 3
Other: Head ultrasound — In cohort 3, a head ultrasound will be carried in addition to the current medical practice.
  This exam is part of current medical practice for other groups.
  Groups: Cohort 3

SUMMARY:
The Zika epidemic has spread into the three French Overseas Departments in the Caribbean (DFAs). It is therefore urgent to set up tools to collect clinical and paraclinical data for the evaluation of potential complications due to having ZIKV infection during pregnancy.

This study is meant to collect, within usual care practices, clinical and paraclinical information (including imaging and laboratory results) as well as biological samples allowing the precise description of the consequences of ZIKV infection during pregnancy.

This study is the 2nd arm of a global research program in the 3 French Overseas Departments in the Caribbean. It is complementary to the first arm (ZIKA-DFA-FE) consisting in the follow-up of women in the French Overseas Departments who are pregnant during the Zika epidemic period.

The study population is made up of infants born during and up to 9 months after the end of the Zika epidemic period in the French Overseas Departments.

The data and biological specimens collected for this project will be done so through the recommended standard of care which has been put in place considering the ZIKV epidemic in the 3 French Overseas Departments, upholding existing recommendations (profession and/or recommendation from the public health authorities)

DETAILED DESCRIPTION:
At birth (from Day 0 to Day 4):

* Standardized clinical examination by a pediatrician
* Capillary blood sample to do ZIKV serology (in the case that no cord-blood sample was taken at birth) through neonatal heel prick (Guthrie's test)
* Cranial ultrasound
* Screening test for hearing capabilities by auditory evoked potentials
* Fundus of the eye or retinal image capture by RetCam®.

Follow-up from Day 4 to 2 years:

- Clinical examination focusing on neuropsychomotor development at the 2nd, 4th, 9th, 18th and 24th month.

ELIGIBILITY:
Cohort 1:

Inclusion criteria:

1. symptomatic acute infection ZIKV has been confirmed in mother by RT-PCR in blood or urine or serology neutralization or other specific technique that would be validated and become available before the end of the epidemic period OR
2. Mother enrollment in ZIKA DFA FE study (Module 1) OR
3. ZIKA seroconversion documented during pregnancy, especially objectified in the pregnant women's monitoring in the modules 3 and 4 of ZIKA-DFA-FE study AND
4. No birth defects in newborn at birth (see Appendix 5).

Exclusion criteria:

1. premature birth (< 35 weeks amenorrhea)
2. Parents refuse or not able to sign the consent form.

Cohort 2:

Inclusion Criteria:

1. Mother enrollment in ZIKA DFA FE study (Module 2) OR
2. Children born from mothers enrolled in ZIKA-DFA-FE study (modules 3 and 4) and having congenital abnormalities discovered at birth

And having at least one of these following abnormalities:

Head circumference (HC) < 2 SD, using Intergrowth curves:

(http://intergrowth21.ndog.ox.ac.uk/Newborn/en/ManualEntry) Presence of birth defects in newborn at birth (see Annex 5)

Exclusion criteria:

1. premature birth (< 35 weeks amenorrhea)
2. Parents refuse or not able to sign the consent form.

Cohort 3:

Inclusion Criteria:

1. Mother enrollment in ZIKA DFA FE study (Module 3 &4)
2. Mother's ZIKV seronegative in childbirth
3. No birth defects in newborn at birth (see Appendix 5).

Exclusion criteria:

1. premature birth (< 35 weeks amenorrhea)
2. Parents refuse or not able to sign the consent form

Ages: 0 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies born during and up to 9 months after the end of the epidemic of ZIKV within the french indies and Guyana.
  3 groups : babies without any congenital abnormalities from mother with ZIKV infection, biologicaly confirmed during the pregnancy (cohort1); babies with congenital abnormalities at birth (cohort 2); babies without any congenital abnormalities from mother without ZIKV infection during the pregnancy (cohort 3)
Sampling Method: Non-Probability Sample
Enrollment: 1180 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Embryofoetopathy incidence within cohort 1 and 3 | 24 months
  incidence comparison between the 2 groups and the calcul of adjusted incidence ratios
Comparison of congenital abnormality incidence rates between cohorts 1 and 3 | 24 months
  * Whether or not the mother was symptomatic for ZIKV infection during pregnancy
  * Gestational age at the moment of ZIKV infection
  * The level of ZIKV viremia at the moment of acute ZIKV infection

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Hoen, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Olivier Flechelles, Principal Investigator — CHU de la Martinique
Locations (6):
- France (6):
  - CH de la Basse Terre, Basse-terre Cedex
  - CH Andrée Rosemon (CHAR), Cayenne Cedex
  - CHU de Martinique, FORT de France Cedex
  - CHU de Pointe à Pitre/Les Abymes, Pointe à Pitre
  - CH de l'Ouest Guyanais Franck Joly (CHOG), Saint-laurent-du-maroni
  - CH LC Fleming, Saint-Martin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grant R, Flechelles O, Tressieres B, Dialo M, Elenga N, Mediamolle N, Mallard A, Hebert JC, Lachaume N, Couchy E, Hoen B, Fontanet A. In utero Zika virus exposure and neurodevelopment at 24 months in toddlers normocephalic at birth: a cohort study. BMC Med. 2021 Jan 21;19(1):12. doi: 10.1186/s12916-020-01888-0. PMID 33472606